CLINICAL TRIAL: NCT06024460
Title: Comparative Effectiveness of Non-pharmacological Treatment and Pharmacological Treatment for Non-acute Lumbar Disc Herniation: a Multi-centered, Pragmatic Randomized Controlled, Parallel-grouped Study
Brief Title: Non-pharmacological Treatment vs Pharmacological Treatment for Non-acute Lumbar Disc Herniation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2023-02
Record Dates: First submitted 2023-07-20; First posted 2023-09-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: The interventional study model in this study is a pragmatic, multi-centered, randomized controlled, parallel-grouped design. This means that the study will involve multiple centers, random assignment of participants into different treatment groups (non-pharmacological treatment arm and pharmacological treatment arm), and a parallel-grouped comparison of the effectiveness of the interventions. The study aims to assess the real-world effectiveness of the treatment strategies in a pragmatic setting, allowing flexibility in treatment decisions based on clinical judgment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-pharmacological treatment strategy (Experimental): Interventions: Non-pharmacological treatment include acupuncture, electroacupuncture, spinal manual therapy, and motion style acupuncture treatment.
  Frequency: Not specified (Twice a week recommended) Duration: Eight weeks.
  Interventions: Procedure: non-pharmacological treatment strategy
- Pharmacological treatment strategy (Active Comparator): Interventions: Active pharmacological treatment involving prescription medication, injection therapy, or other pharmacological interventions.
  Frequency: Not specified (Twice a week recommended) Duration: Eight weeks.
  Interventions: Procedure: pharmacological treatment strategy

INTERVENTIONS:
Procedure: non-pharmacological treatment strategy — Acupuncture, elctroacupuncture, spinal manual therapy, motion style acupucnture treatment
  Arms: Non-pharmacological treatment strategy
Procedure: pharmacological treatment strategy — Prescription medication, injection therapy, nerve blocks, or other pharmacological interventions commonly used for managing lumbar disc herniation.
  This group is treated using the above treatment strategies, and no drug is specified.
  Arms: Pharmacological treatment strategy

SUMMARY:
This is a randomized controlled study comparing non-pharmacological treatment to proactive pharmacological treatment for patient with non-acute lumbar disc herniation with moderate or higher levels of pain. The study involves 200 adult patients aged 19-69, with 50 patients from each participating hospital. Patients will be randomly assigned to either the non-pharmacological treatment group or the pharmacological treatment group 1:1 ratio. Specific interventions will be determined by doctors and Korean medicine doctors without predefined treatment strategies. The non-pharmacological treatment include acupuncture, electroacupuncture, spinal manual therapy and motion style acupuncture. The pharmacological treatment include medication prescription, injection, and nerve block. Treatment period is 8 weeks, and f/u for 3 years.

DETAILED DESCRIPTION:
This is a pragmatic, multi-centered, randomized controlled, parallel-grouped study aiming to compare the effectiveness of a non-pharmacological treatment strategy and a active pharmacological treatment strategy in managing non-acute lumbar disc herniation with moderate or higher levels of pain persisting for more than one month in adult men and women aged 19 to 69 years.

The study will include 200 patients with lumbar disc herniation, with 50 patients from each of the participating hospitals (Jaseng Hospital of Korean Medicine, Daejeon Jaseng Hospital of Korean Medicine, Bucheon Jaseng Hospital of Korean Medicine, Haeundae Jaseng Hospital of Korean Medicine, competitively recruited). The patients will be assigned in a 1:1 ratio to receive either non-pharmacological treatment (100 patients) or active pharmacological treatment (100 patients) in a pragmatic randomized controlled design. The specific interventions for each group will be determined based on clinical judgment by the doctors and Korean medicine doctors involved in the study, without predefining the treatment strategies. The treatment methods, including acupuncture, electroacupuncture, spinal maunal therapy and motion style acupuncture, will be recorded in the case report form for comparative analysis.

For the non-pharmacological treatment group, patients will be recommended to receive non-pharmacological treatment based on TKM. The frequency and specifics of the treatment will be determined by the clinical judgment of the doctors and Korean medicine doctors based on the patient's symptoms, MRI images, and clinical improvement. The treatment will be conducted twice a week for a total of eight weeks, but the frequency may be adjusted according to the patient's condition. Concurrent therapies and adjuvant therapies can be freely chosen by the patients, and the details will be recorded in the case report form.

For the pharmacological treatment group, patients will be educated about proactive pharmacological treatment and recommended to receive pharmacological treatment. The specific pharmacological interventions, such as prescription medication, injection therapy, and nerve block, will be determined by the doctors based on the patient's symptoms, imaging results, and clinical judgment. The details of the prescribed medication, dosage, administration route, and duration will be recorded in the case report form. Similar to the non-pharmacological treatment group, concurrent therapies and adjuvant therapies can be chosen by the patients, and the details will be recorded.

The treatment frequency for the pharmacological treatment group will also be twice a week for a total of eight weeks, with adjustments based on the patient's condition. The effectiveness of the treatment strategies will be assessed through weekly evaluations of the patients' symptoms and treatment progress.

It should be noted that patients are not obligated to strictly follow the assigned treatment strategy, as this is a study recommending a particular treatment strategy rather than enforcing it as a protocol violation.

ELIGIBILITY:
Inclusion Criteria:

* aged 19 to 69 years.
* lower back pain that has persisted for at least 1 month.
* a Numeric Rating Scale (NRS) score of 5 or higher for either lower back pain or radiating leg pain over the past three consecutive days.
* confirmed lumbar disc herniation on MRI that can explain the lower back pain.
* who have provided written informed consent and agreed to participate in the clinical study.

Exclusion Criteria:

* diagnosed with specific severe diseases that could be the cause of lower back pain or leg pain (e.g., spinal metastasis, acute fractures, and spinal dislocation).
* showing progressive neurological deficits or severe neurological symptoms.
* with pain originating from soft tissue disorders other than the spine (e.g., tumors, fibromyalgia, rheumatoid arthritis, gout).
* with other chronic conditions (e.g., stroke and myocardial infarction, renal disease, diabetic neuropathy, dementia, epilepsy) that may interfere with the treatment effect or result interpretation.
* taking steroids, immunosuppressive drugs, psychiatric medications, or other medications that may impact the study results.
* acupuncture or nerve block treatment is inappropriate or unsafe, such as those with a history of bleeding disorders, receiving anticoagulant therapy, or diagnosed with uncontrolled diabetes.
* taken non-steroidal anti-inflammatory drugs (NSAIDs) or other pain-affecting drugs or received acupuncture treatment within the past 5 days.
* Pregnant women, those planning pregnancy, or breastfeeding women.
* within 3 months after lumbar surgery.
* who have not completed participation in another clinical study within the past month or have plans to participate in another clinical study within 6 months from the selection date or during the study participation and follow-up period.

Inability to provide written informed consent.

- Other cases where the researchers determine that participation in the clinical study would be difficult.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Week 1, 5, 9, 13, 26, 39, 52, Month 18, 24, 36
  The Oswestry Disability Index (ODI) is a questionnaire used to assess the functional status and degree of disability caused by lower back pain. It consists of 10 items that evaluate various aspects of daily activities and mobility. Each item is rated on a 6-point scale, with higher scores indicating a greater level of disability.
  From 0 to 100. Higher scores mean a worse outcome.
Numeric Rating Scale for Pain of Dominant Change (NRS for DC) | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 13, 26, 39, 52, Month 18, 24, 36
  The study will evaluate the intensity of lower back pain and radiating leg pain using the Numeric Rating Scale (NRS). Patients will rate their pain levels on a scale from 0 to 10, where 0 represents no pain and 10 represents the most severe imaginable pain. The NRS for Dominant Change (NRS-DC) will be calculated as the higher value between the change in NRS scores from baseline for lower back pain and radiating leg pain. The NRS-DC will serve as a key evaluation indicator for pain intensity.

SECONDARY OUTCOMES:
Recurrence | Week 13, 26, 39, 52, Month 18, 24, 36
  This study will confirm the recurrence of symptoms in patients through a yes or no response.
Numeric Rating Scale (NRS) for Low Back Pain | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 13, 26, 39, 52, Month 18, 24, 36
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participants are asked to report their low back pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable.
Patient Global Impression of Change (PGIC) | Week 9, 13, 26, 39, 52, Month 18, 24, 36
  Participants rate the improvement after treatment on a 7-point Likert scale (1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.)
Fear-Avoidance Beliefs Questionnaire (FABQ) | Week 1, 5, 9, 13, 26, 39, 52, Month 18, 24, 36
  The fear-avoidance belief questionnaire (FABQ) is a questionnaire based on the fear-avoidance model of exaggerated pain perception. The FABQ measures patient's fear of pain and consequent avoidance of physical activity (PA) because of their fear.
  Minimum 0 to maximum 66 scores. Higher score means a worse outcome.
Short Form-12 Health Survey version 2 (SF-12 v2) | Week 1, 5, 9, 13, 26, 39, 52, Month 18, 24, 36
  The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
  Ranging from 0 to 100, higher score means a better outcome.
EuroQol-5 Dimension (EQ-5D-5L) | Week 1, 5, 9, 13, 26, 39, 52, Month 18, 24, 36
  The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about) Ranging from 0 to 1, higher score means a better outcome.
Credibility and Expectancy | Baseline
  The study will measure the level of trust and expectation regarding the effectiveness of the treatment through two questions:
  On a scale from 0 to 10, how much do you believe that traditional herbal medicine treatment will alleviate your symptoms? On a scale from 0 to 10, how much do you believe that drug therapy will alleviate your symptoms? 0 indicates no belief or expectation, and 10 indicates full belief and high expectation.
Intention to Treat | Week 9
  Evaluate participants' intentions if they are willing to receive non-pharmacological treatment strategies or pharmacological treatment strategies in the future on a scale from 0 to 9. 0 indicates no intention, and 10 indicates full belief and high intention.
Work Productivity and Activity Impairment-Specific Health Problem | Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 13, 26, 39, 52, Month 18, 24, 36
  Productivity loss will be assesed by WPAI-SHP. Through the WPAI questionnaire, the overall work productivity, which is a concept combining absenteesim and presenteeism, as well as employment will be investigated and used as outcomes.
Classification of Disc Degeneration | Week 1, 26, 52, Month 24, 36
  Classify the degree of disc degeneration based on the Pfirrmann grading system.
Stages to a Disc Herniation | Week 1, 26, 52, Month 24, 36
  Classify the stage of disc herniation as bulging, protrusion, extrusion, or sequestration/migration.
Herniated Disc Areas | Week 1, 26, 52, Month 24, 36
  Measure the area of the most significant transverse plane slice of the herniated disc on MRI.
Cost Data Survey | Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 13, 26, 39, 52, Month 18, 24, 36
  Measure various cost items related to the treatment, including medical costs, non-medical costs, time costs, and productivity loss costs.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Dr, Study Director — Jaseng Medical Foundation
Locations (4):
- South Korea (4):
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi-do
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim D, Lee YJ, Yang C, Ahn YJ, Kim S, Lee Y, Cho HW, Han CH, Ha IH. Non-Pharmacological and Pharmacological Treatments for Non-Acute Lumbar Disc Herniation: A Protocol for a Multicenter Pragmatic Trial. J Pain Res. 2025 Dec 26;18:7167-7178. doi: 10.2147/JPR.S568386. eCollection 2025. PMID 41477591